CLINICAL TRIAL: NCT02388815
Title: Evaluation of the Accuracy of the Abbott Sensor Based Glucose Monitoring System - Paediatric Label Extension Study (CE)
Brief Title: Abbott Sensor Based Glucose Monitoring System Paediatric Study
Acronym: BEAGLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ADC-UK-VAL-14022
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Results first posted 2016-04-12 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Sensing Technology
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): FreeStyle Libre Flash Glucose Monitoring System
  Interventions: Device: FreeStyle Libre Flash Glucose Monitoring System

INTERVENTIONS:
Device: FreeStyle Libre Flash Glucose Monitoring System — Subjects will wear the Abbott Sensor Based Glucose Monitoring System masked for 14 days.
  During these 14 days subjects will be asked to perform 4 blood glucose tests (meals time and before bedtime) per day. At the same time as the blood glucose test a sensor scan is performed.

SUMMARY:
To evaluate the point accuracy of the Abbott Sensor Based Glucose Monitoring System when used at home by children with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 4 years, ≤17 years
* Each participant has an identified Caregiver of ≥18 years
* Type 1 or type 2 diabetes using insulin administered by injections or continuous subcutaneous insulin infusion (CSII)
* Currently testing blood glucose, on average at least 2 times per day
* In the investigator's opinion, technically capable of using device (participant and/or caregiver).

Exclusion Criteria:

* Concomitant disease or condition that may compromise patient safety including and not limited to; cystic fibrosis, severe mental illness, known or suspected eating disorder or any uncontrolled long term medical condition
* Currently prescribed oral steroid therapy for any acute or chronic condition
* Currently receiving dialysis treatment or planning to receive dialysis during the study
* Female participant known to be pregnant
* Participating in another study of a glucose monitoring device or drug that could affect glucose measurements or management
* Currently using a continuous glucose monitoring (CGM) device
* Known (or suspected) allergy to medical grade adhesives
* In the investigator's opinion the participant or caregiver is unsuitable to participate due to any other cause/reason (both patient and caregiver considered)

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United Kingdom (9):
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Royal Devon and Exeter NHS Foundation Trust, Exeter
  - Harrogate & District NHS Foundation Trust, Harrogate
  - St. James University Hospital, Leeds Teaching Hospitals NHS Trust, Leeds
  - Northampton General Hospital NHS Trust, Northampton
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford Radcliffe Hospital NHS Trust, Oxford
  - Southampton University Hospital NHS Trust, Southampton

REFERENCES:
- [Derived] Edge J, Acerini C, Campbell F, Hamilton-Shield J, Moudiotis C, Rahman S, Randell T, Smith A, Trevelyan N. An alternative sensor-based method for glucose monitoring in children and young people with diabetes. Arch Dis Child. 2017 Jun;102(6):543-549. doi: 10.1136/archdischild-2016-311530. Epub 2017 Jan 30. PMID 28137708

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 89 subjects consented and were enrolled into the study.
Period: Overall Study
Arm/Group | FreeStyle Libre Flash Glucose Monitoring System
Started | 89
Completed | 85
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | FreeStyle Libre Flash Glucose Monitoring System
Number analyzed (Participants) | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 89
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 45
Region of Enrollment [Number; unit: participants]
  United Kingdom | 89

OUTCOME MEASURES:

1. Primary Outcome: Point Accuracy
Description: Point accuracy of Sensor based glucose values versus fingerstick blood glucose determined as % within Consensus Error Grid zone A.
  The Consensus Error Grid was developed from a survey of 100 clinicians to evaluate the accuracy of glucose measurements. Glucose results from the system under test (y) are paired with those from a reference method (x) and each (x,y) point is plotted on a grid. The grid has 5 risk categories, assigned by the clinicians surveyed. Risk categories (in order of increasing severity) are: Zone A: no effect on clinical action; Zone B: altered clinical action or little or no effect on clinical outcome; Zone C: altered clinical action likely to effect clinical outcome; Zone D: altered clinical action, could have significant medical risk; Zone E: altered clinical action, could have dangerous consequences.
  Result were calculated for all subjects ie total number of sensor results and fingerstick blood glucose results divided by the total number of results x 100.
Time Frame: 14 days
Population: One subject withdrew prior to having a sensor applied, another did not perform any blood glucose tests on the FreeStyle Libre. Neither subject could be included in the accuracy analysis, both are included in the safety analysis.
Measure: Number (95% Confidence Interval); unit: percentage of glucose results in zone A
Arm/Group | FreeStyle Libre Flash Glucose Monitoring System
Number analyzed (Participants) | 87
percentage of glucose results in zone A | 83.8 [82.5 to 86.3]

ADVERSE EVENTS:
Time Frame: Adverse Events collected from enrolment to completion by last subject (2.5 months)
Arm/Group | FreeStyle Libre Flash Glucose Monitoring System
Serious Adverse Events (participants affected / at risk) | 1/89
Other Adverse Events (participants affected / at risk) | 15/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FreeStyle Libre Flash Glucose Monitoring System (N=89)
Painful right leg (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FreeStyle Libre Flash Glucose Monitoring System (N=89)
Common cold (General disorders) | 9 (9)
Headache (General disorders) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days